CLINICAL TRIAL: NCT04071080
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study of Oral Fluorescite to Confirm the Authenticity of Point of Care Urine Samples
Brief Title: The Study of Oral Fluorescite to Confirm the Authenticity of Point of Care Urine Samples
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UpTru Inc. (Industry)
Collaborators: Medicor Research Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: PH1.20180001
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Urine Sample Authenticity
MeSH Terms: interventions — Fluorescein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 100mg Fluorescein disodium (Experimental): 100mg Fluorescein disodium will be mixed with 500mL of Gatorade and taken orally by the participant
  Interventions: Drug: fluorescein sodium
- Placebo (Placebo Comparator): 500mL of Gatorade taken orally by the participant
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fluorescein sodium — Fluorescein sodium in 500mL Gatorade
  Other Names: Fluorescite
  Arms: 100mg Fluorescein disodium
Drug: Placebo — 500mL Gatorade
  Arms: Placebo

SUMMARY:
During this study, participants will ingest 100 mg of fluorescein disodium or a placebo (no drug) mixed in GatoradeTM. Participants will then provide a urine sample after 10, 15, 20 or 30 minutes to see if the investigator can detect fluorescein fluorescence (light) in the urine.

DETAILED DESCRIPTION:
Every year, millions of dollars are spent on urine drug testing. Urine samples are generally provided in an unwitnessed fashion. Only a small percentage of samples involve direct observation of urination. The authenticity of the provided sample greatly affects its clinical utility and/or the validity of the test results. Direct observation of urination can be unpleasant and humiliating for people. For the institution, there are increased costs (for example, staff, insurance) and risks regarding impropriety when direct observation is utilized.

Participants are being asked to take part in a research study of an approved drug called FluoresciteTM. FluoresciteTM is an intravenous drug (administered into a vein) that has been approved by Health Canada. The active ingredient in FluoresciteTM is fluorescein disodium (10% fluorescein disodium in sterile water).

Fluorescein disodium has been used medically for over fifty years. It is a fluorophore (emits light, similar to a yellow glowstick) that is most commonly used in ophthalmology (the study and treatment of disorders and diseases of the eye). It is currently used in angiography (to view blood vessels), or topically for staining the eye's cornea. FluoresciteTM or fluorescein disodium has not been approved by Health Canada for oral administration.

During this study, participants will ingest 100 mg of fluorescein disodium or a placebo (no drug) mixed in GatoradeTM. The Investigator will then ask the participant to provide a urine sample after 10, 15, 20 or 30 minutes to see if he can detect fluorescence (light) in the urine.

The purpose of this study is to:

* Develop a new standardized protocol for urine sampling that will increase sample authenticity and make the situation between the patient/physician more pleasant.
* To evaluate the safety and tolerability of orally ingested fluorescein disodium.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to comply with visits and study procedures.
* Healthy males and females between the age of 18 and 55.
* Female subjects are eligible to participate if they are not pregnant, breastfeeding and at least one of the following conditions apply:

  * Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective (based on the investigator's judgment) for 28 days before/after study drug administration.
  * Is not of WOCBP (Postmenopausal and/or surgically sterile)
* Male subjects must use effective birth control methods and must not donate sperm until 2 weeks after treatment.

Exclusion Criteria:

* Staff members involved in the conduct of the study or their family members or site staff members supervised by the investigator. Subjects who are UPTru or Medicor employees, including their family members, directly involved in the conduct of the study are also not eligible to participate.
* Participants involved in any other study using an investigational product within 30 days or 5 half-lives (if known) prior to screening.
* Participants with any history of the following conditions:

  * Known history of allergy (such as food or drug-induced urticaria, asthma, eczema or allergic rhinitis) or known allergy to fluorescein disodium or any component of FluoresciteTM or GatoradeTM.
  * Jaundice, bronchial asthma, cirrhosis, uncontrolled diabetes (HbA1c ≥ 7.0), renal failure (calculated creatinine clearance of < 35 mL/min), cancer, HIV or hepatitis B/C.
* Participants with a life expectancy of fewer than 5 years.
* In the opinion of the investigator, any clinically significant abnormal ECG, vitals or laboratory result during screening that could put the participant at risk or affect the results of the study.
* Any concomitant medication that could potentially interact with the study drug or affect the results of the study (based on the investigator's opinion).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with detectable urine fluorescence using an ophtalmoscope equipped with a cobalt blue filter | Up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medicor Research Inc., Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No